CLINICAL TRIAL: NCT07257341
Title: Pilot Study of Normative Range of Field of Binocular Single Vision in Adults in Singapore
Acronym: NORVIBAS
Status: Recruiting | Type: Observational
Sponsor: Tan Tock Seng Hospital (Other)
Responsible Party: Principal Investigator, Daniel Chin Yuxiang, Associate Consultant, Tan Tock Seng Hospital
Other Study IDs: 2025-1293
Record Dates: First submitted 2025-11-20; First posted 2025-12-02 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Binocular Visual Function
Keywords: Binocular field of vision

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Field of Binocular Single Vision — The intervention involves a single field of binocular single vision assessment using the Takagi MT-325UD Projection Perimeter. Participants undergo binocular testing where they fixate and follow a single round light stimulus as it moves throughout the perimeter bowl. When participants perceive two distinct light stimuli (indicating loss of binocular single vision), they press a buzzer. The orthoptist records these responses and plots the boundaries on a standardised recording sheet to map the participant's field of binocular single vision.
  This intervention addresses significant limitations of the current gold standard established by Feibel & Roper-Hall (1974). The original study was conducted with "several" normal individuals (likely fewer than 10 participants) of Caucasian descent in St Louis, Missouri, creating potential issues with statistical power and population applicability. Our study uses a larger, more robust sample size of 32 participants specifically from Singapore's Asian

SUMMARY:
The assessment and monitoring of the field of binocular single vision remains a crucial aspect of ophthalmological care, yet current clinical practice relies on normative standards established by Feibel & Roper-Hall in 1974 that present significant limitations for contemporary application. The original study, conducted with a demographically homogeneous Caucasian population in St Louis using only "several" normal individuals, raises concerns regarding its applicability to Asian populations, particularly in Singapore, where ethnic and genetic factors may influence ocular characteristics. The limited sample size significantly increases the likelihood of Type II errors, whilst the temporal gap of over five decades introduces additional concerns regarding population changes, environmental factors, and advances in measurement techniques that have not been incorporated into current normative data. Given these substantial limitations in demographic representation, statistical power, and temporal relevance, there exists a pressing need to establish population-specific normative data for the field of binocular single vision in Singapore's adult population, which would provide more clinically relevant reference values and potentially improve diagnostic accuracy for ocular conditions in the local context.

DETAILED DESCRIPTION:
The assessment and monitoring of the field of binocular single vision is a crucial aspect of ophthalmological care, particularly in the management of oculoplastics and strabismus. Currently, clinicians worldwide, including those in Singapore, rely on the normal boundary of the field of binocular single vision established by Doctor Robert M. Feibel & Gill Roper-Hall in 1974 as the gold-standard parameter for clinical assessment. However, this long-standing standard raises several significant concerns regarding its applicability to our current population.

The original study by Feibel & Roper-Hall was conducted in St Louis, Missouri, United States of America, with participants who were likely of Caucasian descent. This demographic composition presents a potential limitation when applying these standards to Asian populations, particularly in Singapore, where ethnic and genetic factors may influence ocular characteristics. Furthermore, the study's methodology involved only "several" normal individuals, suggesting a sample size of more than two but fewer than ten participants. A sample size of this limited scope significantly increases the likelihood of Type II errors, potentially compromising the statistical power and reliability of the established normative values.

The temporal gap of over five decades since the original study adds another layer of concern. Population characteristics, environmental factors, and lifestyle patterns have undergone substantial changes during this period, potentially affecting ocular health parameters. Additionally, advances in measurement techniques and an understanding of ocular physiology suggest the need for updated normative data that reflect current population characteristics and incorporate modern assessment methodologies.

Given these limitations, there is a pressing need to establish population-specific normative data for the field of binocular single vision in Singapore's adult population. This would not only provide more relevant reference values for clinical assessment but also potentially improve the accuracy of diagnosis and monitoring of various ocular conditions in our local context.

ELIGIBILITY:
Inclusion Criteria:

* Age: 21 to 59 years old
* Gender: Males or females
* Ethnicity: Asian descent.
* Language comprehension: Able to understand verbal spoken instructions in:

  • British/American English
  * Mandarin Chinese
  * Bahasa Melayu
* Protocol compliance: Ability to comply with the study protocol, as determined by the investigator's judgment
* Consent capacity: Must be able to understand and provide informed consent, with signed informed consent form required before any study assessments

Exclusion Criteria:

- Communication barrier: Unable to understand verbal spoken instructions

* Medical history:

  * Any facial trauma
  * Any ocular trauma
  * Any head trauma
  * Any history of ocular disease
  * Any history of ocular surgery
  * Systemic condition(s)
* Near visual acuity:

  o Right eye & Left eye monocularly, binocularly unaided near vision: worse than N6 at 40cm from participant's nose
* Ocular alignment:

  o Prism cover test at near (30cm) of equal or greater than 10 prism diopters at these positions of gaze:
  * Primary gaze
  * Right gaze
  * Left gaze
  * Up gaze
  * Down gaze
* Extraocular movement:

  o Extraocular movement of over-action or under-action of equal or greater than 0.5 in any of the nine cardinal positions of gaze
* Confrontational Visual field:

  o Abnormal monocular visual field on confrontational visual field test
* Hess chart test o Abnormal or asymmetry in pattern of extraocular muscle action in Hess chart test

Ages: 21 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy Individuals
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-10-15 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-10-14 (Estimated)

PRIMARY OUTCOMES:
Field of Binocular Single Vision in Asian population | up to 20 minutes during 1 study visit.
  Establish comprehensive normative range of field of binocular single vision (BSV) specifically for healthy adults in Singapore's population aged 21-59, creating locally relevant reference standards that reflect ethnic, genetic, and contemporary population.
  BSV is the ability to use both eyes simultaneously and coordinate the slightly different images from each eye into a single, unified, three-dimensional mental percept. The "field of binocular single vision" is the specific area within the overall visual field where this fusion and single vision can be maintained.
  To measure the field of BSV using Goldmann perimetry, a moving light stimulus is presented while the patient uses both eyes. The test maps the area where the patient can maintain fusion (single vision). The boundary where fusion breaks (and diplopia starts) is plotted across different directions to define the BSV field.

SECONDARY OUTCOMES:
Comparison of current field of binocular single vision gold standard between Caucasian population vs Asian population | Up to 20 minutes during 1 study visit.
  Conduct rigorous statistical comparison between newly established Singapore normative values and existing Feibel & Roper-Hall (1974) standards to quantify differences and determine clinical significance.
  Current benchmarks are based on a 1974 U.S. study by Feibel & Roper-Hall that involved fewer than ten Caucasian subjects and no Asian representation. Consequently, clinicians may over- or under-diagnose ocular deviation and fusion deficits in Asian patients. The study validates a modern methodology using the Takagi MT-325UD Projection Perimeter to map BSV fields under standardized conditions.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Chin, MBBS, Principal Investigator — Tan Tock Seng Hospital; Sebastian Yue, MSc, Study Director — Tan Tock Seng Hospital
Locations (1):
- Tan Tock Seng Hospital, Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No
Participant data cannot be shared due to local governing laws and institutional regulations.

REFERENCES:
- [Result] Feibel RM, Roper-Hall G. Evaluation of the field of binocular single vision in incomitant strabismus. Am J Ophthalmol. 1974 Nov;78(5):800-5. doi: 10.1016/0002-9394(74)90303-1. No abstract available. PMID 4425006
- [Result] Kakizaki H, Umezawa N, Takahashi Y, Selva D. Binocular single vision field. Ophthalmology. 2009 Feb;116(2):364. doi: 10.1016/j.ophtha.2008.08.046. No abstract available. PMID 19187829

DOCUMENTS (1):
  • Study Protocol (2025-12-15): https://cdn.clinicaltrials.gov/large-docs/41/NCT07257341/Prot_001.pdf